CLINICAL TRIAL: NCT04161391
Title: A Phase 1/2 Study of TPX-0046, A Novel Oral RET/SRC Inhibitor in Adult Subjects With Advanced/Metastatic Solid Tumors Harboring Oncogenic RET Fusions or Mutations
Brief Title: Study of TPX-0046, A RET/SRC Inhibitor in Adult Subjects With Advanced Solid Tumors Harboring RET Fusions or Mutations
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Adverse change in the risk/benefit.
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA129-1036; CA129-1036 (Other: Bristol-Myers Squibb Protocol ID); TPX-0046-01 (Other: Turning Point Therapeutics Protocol ID)
Record Dates: First submitted 2019-11-11; First posted 2019-11-13 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer; Medullary Thyroid Cancer; RET Gene Mutation; Metastatic Solid Tumor; Advanced Solid Tumor
Keywords: Non small cell lung cancer; Non-small cell lung cancer; NSCLC; Medullary Thyroid Cancer; MTC; RET gene mutation; RET gene alteration; Advanced non small cell lung cancer; Advanced/metastatic disease; lung cancer; lung adenocarcinoma; Metastatic solid tumor; Advanced Solid Tumors; RET gene fusion; RET inhibitor; SRC; TPX-0046; Thyroid cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Medullary; Neoplasm Metastasis; Lung Neoplasms; Adenocarcinoma of Lung; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TPX-0046 (Experimental): The Phase 1 part of the study will determine the safety, tolerability, PK, MTD, and RP2D of TPX-0046.
  The food-effect sub-study determines the effect of food on a dose of TPX-0046 at the RP2D dose level.
  The Phase 2 part of the study will determine the safety, tolerability, PK, and preliminary efficacy in specific cohorts.
  Phase 2 Cohorts:
  * Cohort I (NSCLC + RET fusion, RET TKI Therapy Naive)
  * Cohort II (NSCLC + RET fusion, RET TKI Therapy Pre-treated)
  * Cohort III (MTC + RET mutation, RET TKI Therapy Naive)
  * Cohort IV (MTC + RET mutation, RET TKI Therapy Pre-treated)
  * Cohort V (advanced/metastatic tumor with RET fusion or mutation, RET TKI Therapy Naive)
  * Cohort VI (advanced/metastatic tumor with RET fusion or mutation, RET TKI Therapy Pre-Treated)
  Interventions: Drug: TPX-0046

INTERVENTIONS:
Drug: TPX-0046 — Oral TPX-0046 capsules

SUMMARY:
A phase 1/2, first-in-human, open-label study to determine the safety, tolerability, PK, and preliminary efficacy of the novel RET/SRC inhibitor TPX-0046 in adult subjects with advanced or metastatic solid tumors harboring RET mutations or alterations. The study consists of three portions: 1) Phase 1 Dose Escalation and Food Effect Sub-study, and 2) Phase 1 dose expansion and 3) Phase 2 efficacy evaluation.

DETAILED DESCRIPTION:
Phase 1 Dose Escalation and Dose Expansion: To evaluate the overall safety profile, characterize the PK profiles and assess the preliminary efficacy of TPX-0046 in adults subjects with advanced solid tumors harboring oncogenic RET fusions or mutations.

Food Effect Sub-Study: To determine the effect of food on PK of TPX-0046 in adult subjects with advanced or metastatic solid tumors harboring oncogenic RET fusions or mutations.

Phase 2 Efficacy Evaluation: To determine the overall safety and anti-tumor efficacy of TPX-0046 in defined cohorts of subjects with advanced/metastatic solid tumors harboring oncogenic RET fusions or mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 (or age ≥ 20 as required by local regulation).
2. Histological or cytological confirmation of advanced/metastatic solid tumors harboring oncogenic RET fusions or mutations, who either have disease progression on, or are intolerant to standard therapy; OR are ineligible for standard therapy or for whom no standard therapy exists; OR are unlikely to tolerate or derive clinical benefit from standard therapy in the opinion of the Investigator OR have declined standard therapy.
3. ECOG performance status ≤ 1.
4. Existence of measurable or evaluable disease (according to Response evaluation criteria in solid tumors [RECIST v1.1] criteria).
5. Subjects with asymptomatic primary CNS tumors or brain metastases are eligible for the study if they meet protocol specified criteria.
6. Adequate organ function.
7. Life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Locally advanced solid tumor that is a candidate for curative treatment through radical surgery and/or radiotherapy, or chemotherapy.
2. Presence or history of any other primary malignancy within 3 years other than a history of adequately treated basal or squamous cell carcinoma of the skin, or any adequately treated in situ carcinoma.
3. Major surgery within four weeks of the start of therapy.
4. Clinically significant cardiovascular disease (either active or within six months before enrollment): myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association Classification Class ≥ II), cerebrovascular accident or transient ischemic attack, symptomatic bradycardia, requirement for anti-arrhythmic medication. Ongoing cardiac dysrhythmias of CTCAE version 5.0 grade ≥ 2.
5. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (ECG interval measured from the onset of the QRS complex to the end of the T wave) for heart rate (QTc) > 470 msec obtained from three ECGs, using the screening clinic ECG machine-derived QTc value
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec)
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication known to prolong the QT interval
6. Known clinically significant active infections not controlled with systemic treatment (bacterial, fungal, viral including HIV positivity).
7. Gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact drug absorption.
8. Subjects being treated with or anticipating the need for treatment with strong CYP3A4 inhibitors or inducers.
9. Subjects with current or anticipated need for drugs that are sensitive CYP2C9 substrates with narrow therapeutic indices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (20):
  - Local Institution - 2129, La Jolla, California
  - Local Institution - 2128, Orange, California
  - Local Institution - 2122, Aurora, Colorado
  - SCRI - HealthOne Denver, Denver, Colorado
  - Local Institution - 2126, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Local Institution - 2130, Tampa, Florida
  - Local Institution - 2127, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Local Institution - 2124, Ann Arbor, Michigan
  - Local Institution - 2131, Detroit, Michigan
  - Mayo Clinic - Arizona, Rochester, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 2137, Philadelphia, Pennsylvania
  - Local Institution - 2120, Houston, Texas
  - Baylor College of Medicine - Baylor Heart Clinic, Houston, Texas
  - Local Institution - 2135, Fairfax, Virginia
  - Local Institution - 2132, Seattle, Washington
- Local Institution - 6320, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg QD: TPX-0046 10 mg daily (QD) in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
- 10 mg BID: TPX-0046 10 mg twice a day (BID) in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
- 20 mg QD: TPX-0046 20 mg daily (QD) in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
- 30 mg QD: TPX-0046 30 mg daily (QD) in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
- 20 mg BID: TPX-0046 20 mg twice a day (BID) in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
- 20 mg QD to 30 mg QD: TPX-0046 20 mg daily (QD) for the first 14 days, then 30 mg daily in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
- 20 mg QD to 20 mg BID: TPX-0046 20 mg daily (QD) for the first 14 days, then 40 mg in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
- 20 mg QD to 40 mg QD: TPX-0046 20 mg (daily) QD for the first 14 days, then 40 mg in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
- 10 mg QD to 10 mg BID: TPX-0046 10 mg daily (QD) for the first 14 days, then 20 mg in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
Period: Overall Study
Arm/Group | 10 mg QD | 10 mg BID | 20 mg QD | 30 mg QD | 20 mg BID | 20 mg QD to 30 mg QD | 20 mg QD to 20 mg BID | 20 mg QD to 40 mg QD | 10 mg QD to 10 mg BID
Started | 4 | 4 | 4 | 8 | 3 | 3 | 7 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 4 | 8 | 3 | 3 | 7 | 6 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0
Not completed — Progressive Disease | 4 | 3 | 3 | 5 | 3 | 3 | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg QD | 10 mg BID | 20 mg QD | 30 mg QD | 20 mg BID | 20 mg QD to 30 mg QD | 20 mg QD to 20 mg BID | 20 mg QD to 40 mg QD | 10 mg QD to 10 mg BID | Total
Number analyzed (Participants) | 4 | 4 | 4 | 8 | 3 | 3 | 7 | 6 | 2 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (5.97) | 58.0 (10.23) | 60.8 (3.59) | 60.1 (15.69) | 59.3 (19.50) | 64.7 (9.45) | 62.7 (10.36) | 60.5 (8.87) | 61.5 (12.02) | 60.8 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 5 | 0 | 1 | 5 | 2 | 1 | 18
  Male | 3 | 2 | 3 | 3 | 3 | 2 | 2 | 4 | 1 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 2 | 3 | 3 | 7 | 2 | 3 | 7 | 5 | 2 | 34
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 1 | 3 | 4 | 5 | 2 | 3 | 7 | 3 | 0 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) of TPX-0046
Description: Participants are eligible for DLT evaluation if they experience a DLT after at least one dose of TPX-0046, or do not experience a DLT after taking at least 75% of the doses expected during the DLT evaluation period. Some adverse events, graded using Common Terminology for Adverse Events (CTCAE) v. 5.0, for defining DLTs include:
  * Toxicities resulting in an excessive number of missed doses;
  * Hematologic: CTCAE grade ≥ 4 neutropenia, CTCAE grade ≥ 4 platelet count decrease, CTCAE grade ≥ 4 anemia, CTCAE grade ≥ 3 febrile neutropenia;
  * Renal: CTCAE grade ≥ 3 creatinine increase;
  * Hepatic: CTCAE grade ≥ 3 total bilirubin elevation;
  * Pancreatic: CTCAE grade 3 serum amylase or lipase increased with clinical symptoms or any grade ≥ serum amylase;
  * Cardiac: CTCAE grade ≥ 3;
  * Other AEs: CTCAE grade 3 vomiting or nausea that does not resolve to grade ≤ 1 within 4 days despite optimal anti-emetic therapy or any grade ≥ 4 vomiting
Time Frame: 28 days following the first highest dose of the dose regimen administered in Cycle 1
Population: DLT evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD | 10 mg BID | 20 mg QD | 30 mg QD | 20 mg QD to 30 mg QD | 20 mg QD to 20 mg BID | 20 mg QD to 40 mg QD | 10 mg QD to 10 mg BID | 20 mg BID
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 2 | 2 | 4 | 1 | 0
Participants | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of TPX-0046
Description: The MTD is defined as the highest dose level of TPX-0046 observed to cause a dose limiting toxicity (DLT) in fewer than 33% of the treated participants in the first treatment cycle (ie, Cycle 1, 28 days).
Time Frame: 28 days following the first highest dose of the dose regimen administered in Cycle 1
Population: All treated participants
Measure: Number; unit: mg
Groups:
- Phase 1 Dose Escalation: TPX-0046 given across 9 dose level cohorts in 28-day continuous cycles until disease progression, unacceptable toxicity, the ability to move to alternative care is identified, or withdrawal of consent
Arm/Group | Phase 1 Dose Escalation
Number analyzed (Participants) | 41
mg | 32.54

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 41 months). SAEs and Other AEs were assessed from first dose to 28 days post the last dose (up to approximately an average of 6 months and a maximum of 27 months).
Arm/Group | 10 mg QD | 10 mg BID | 20 mg QD | 30 mg QD | 20 mg BID | 20 mg QD to 30 mg QD | 20 mg QD to 20 mg BID | 20 mg QD to 40 mg QD | 10 mg QD to 10 mg BID
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/4 | 4/4 | 4/8 | 2/3 | 2/3 | 5/7 | 2/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/4 | 4/4 | 7/8 | 2/3 | 0/3 | 6/7 | 4/6 | 1/2
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 8/8 | 3/3 | 3/3 | 7/7 | 6/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg QD (N=4) | 10 mg BID (N=4) | 20 mg QD (N=4) | 30 mg QD (N=8) | 20 mg BID (N=3) | 20 mg QD to 30 mg QD (N=3) | 20 mg QD to 20 mg BID (N=7) | 20 mg QD to 40 mg QD (N=6) | 10 mg QD to 10 mg BID (N=2)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg QD (N=4) | 10 mg BID (N=4) | 20 mg QD (N=4) | 30 mg QD (N=8) | 20 mg BID (N=3) | 20 mg QD to 30 mg QD (N=3) | 20 mg QD to 20 mg BID (N=7) | 20 mg QD to 40 mg QD (N=6) | 10 mg QD to 10 mg BID (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0
Macular oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Serous retinopathy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 3 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 0 | 1 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 2 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Bacterial test (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cells in urine (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Escherichia test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 2 | 3 | 0 | 1 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary sediment present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine ketone body present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 1 | 0 | 3 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 2 | 2 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 3 | 4 | 0 | 2 | 4 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 3 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
As the study enrollment will close prior to completing Phase 1 dose escalation, the Phase 1 food effect substudy, Phase 1 dose expansion, and Phase 2 activities will not take place.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04161391/Prot_SAP_000.pdf